CLINICAL TRIAL: NCT06865976
Title: Genomic and Proteomic Analysis of Programmed Cell Death Mechanisms in Peri-implant Disease
Brief Title: Genomic and Proteomic Analyses of Apoptosis Mechanisms in Diseased Peri-implant Tissue
Status: Completed | Type: Observational
Sponsor: Sakarya University (Other)
Collaborators: University of Turku (Other); University of Helsinki (Other)
Responsible Party: Principal Investigator, Dogukan Yilmaz, Associate Professor, Sakarya University
Other Study IDs: E-16214662-050.01.04-85,162-21; BIDEB-1059B192100836 (Other Grant/Funding Number: TUBITAK)
Record Dates: First submitted 2025-03-01; First posted 2025-03-10 (Actual); Last update posted 2025-03-10 (Actual); Status verified 2022-06

CONDITIONS: Apoptosis; Apoptosis Regulatory Proteins; Proteases; Peri-Implantitis and Peri-implant Mucositis
MeSH Terms: conditions — Peri-Implantitis

STUDY DESIGN:
Observational Model: Other | Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

GROUPS / COHORTS (3):
- Control: peri-implant tissue health
  Interventions: Procedure: Second stage surgery
- peri-implant mucositis: Peri-implant mucositis was diagnosed in cases of bleeding and/or suppuration upon probing, with no evidence of bone loss beyond the crestal level changes associated with initial bone remodeling, as determined by comparing follow-up and baseline radiographs.
  Interventions: Procedure: Non-Surgical Intervention
- peri-implantitis: Peri-implantitis was diagnosed based on the presence of bleeding and/or suppuration upon probing, probing depths ≥6 mm, and radiographic bone levels ≥3 mm apical to the most coronal portion of the intraosseous part of the dental implant (Berglundh et al., 2018).
  Interventions: Procedure: Surgical peri-implant therapy

INTERVENTIONS:
Procedure: Non-Surgical Intervention — For non-surgical treatment of peri-implant mucositis, granulation tissues were removed by titanium curettes (Hu-Friedy, Titanium Implant Scaler Mini-Five, Chicago, IL, USA) during mechanical debridement under local anesthesia
  Groups: peri-implant mucositis
Procedure: Surgical peri-implant therapy — In cases requiring surgical intervention for peri-implantitis, mucoperiosteal flaps were elevated on both vestibular and oral aspects after administration of local anesthesia (articaine with epinephrine 1:200,000) to expose the peri-implant defect. Granulation tissue from the bony defect area was meticulously excised using by titanium curettes (Hu-Friedy, Titanium Implant Scaler Mini-Five, Chicago, IL, USA).
  Groups: peri-implantitis
Procedure: Second stage surgery — Healthy peri-implant mucosa samples were obtained during the second-stage surgery of implant placement procedures. These samples consisted of incisional biopsies of peri-implant mucosa in direct contact with the implant surface.
  Groups: Control

SUMMARY:
A total of 72 individuals were included in the study: 23 with peri-implant mucositis, 25 with peri-implantitis, and 24 healthy controls. Clinical and radiological parameters, including keratinized mucosa width, modified bleeding index, probing depth, modified plaque index, modified gingival index, and marginal bone loss percentage, were recorded. Granulation tissues were collected during peri-implant disease treatments, while healthy control tissues were obtained during the second stage of implant surgery. Tissue levels of Bcl-2 family pro-apoptotic and anti-apoptotic proteins were measured using multiplex immunoassay, and tissue levels of P. gingivalis gingipain and T. denticola dentilisin with immunoblotting.

DETAILED DESCRIPTION:
The study received ethical approval from the Clinical Research Committee of Sakarya University Faculty of Medicine (Approval number: E-16214662-050.01.04-85,162-217) and was conducted in accordance with the ethical principles outlined in the Declaration of Helsinki. The study protocol was thoroughly explained to all participants, and written informed consent was obtained prior to their inclusion. Recruitment took place between March 2021 and June 2022, involving patients who attended the clinics of the Department of Periodontology, Sakarya University. These patients were either in the maintenance phase following dental implant therapy, actively undergoing implant treatment, or presenting with complications related to dental implants placed at other centers. A total of 72 participants, encompassing 72 dental implants, were enrolled in the study. These participants were categorized as follows: 23 systemically healthy individuals with peri-implant mucositis, 25 individuals with peri-implantitis, and 24 healthy controls. Participant demographics, along with medical and dental histories, were collected during interviews. A comprehensive full-mouth periodontal examination was conducted, and the following clinical parameters were measured at six sites around each implant using a calibrated manual periodontal probe (Hu-Friedy, Chicago, IL, USA): keratinized mucosa width (KTW), modified bleeding index (mBI), probing depth (PD), modified plaque index (mPI), and modified gingival index (mGI). All assessments were performed by a single calibrated periodontist (DY, Kappa coefficient: 0.92). Radiographic evaluations of marginal alveolar bone levels and bone loss percentages were conducted using ImageJ software (ImageJ, Wisconsin, USA). Peri-implant tissue health was classified in accordance with the 2017 classification of Periodontal and Peri-Implant Diseases.

Clinical Procedures and Tissue Sampling Following the baseline assessments, all participants underwent full-mouth prophylaxis and oral hygiene motivation as recommended by EFP treatment guideline. Patients diagnosed with peri-implant mucositis or peri-implantitis were treated by a single periodontist (DY). Granulation tissue samples were collected during the treatment of peri-implant mucositis (non-surgical) and peri-implantitis (resective, reconstructive, or combined surgical approaches). All granulation and mucosal tissue samples were immediately placed into Eppendorf tubes and stored at -80°C. Subsequently, the samples were transported to the Institute of Dentistry, University of Turku and Helsinki University Hospital, University of Helsinki, under dry ice conditions for biochemical analyses. Maintenance therapy was provided to all patients with peri-implant diseases upon completion of their respective treatment protocols.

Analyses of Bcl-2 Family Proteins The thawed tissue samples were first weighed and subsequently sectioned into small pieces with disposable scalpels (#11 and #15, Feather Safety Razor Co., Ltd, Osaka, Japan). The processed tissue fragments were transferred to 2 mL tubes containing four ultrapure zirconium microspheres (3 mm diameter) and 400 μL of lysis buffer. Homogenization was performed using a high-speed tissue homogenizer (TissueLyzer LT, Qiagen, Hilden, Germany) set at 2000 rpm for four cycles of 60 seconds each, with 20 second intervals on ice to prevent overheating. After homogenization, the samples were centrifuged at 10000 rpm for 4 minutes, and the zirconium beads were removed. Ultrasonication (UP50H, Hielscher, Teltow, Germany) was performed at 0.5 cycle and 100% amplitude in three 5-second cycles, with 20-second intervals on ice between the cycles. The samples were then centrifuged again at 10000 rpm for 4 minutes, and the supernatants were carefully transferred to new tubes. Total protein concentrations in the samples were measured by the Bradford assay. The levels of Bcl-2 family proteins were quantified using a bead-based immunoassay system (Luminex xMAP, Luminex Corporation, Austin, TX, USA) with commercially available kits (Bio-Plex Pro RBM Apoptosis Assays, Bio-Rad Laboratories, Hercules, CA, USA) following the manufacturer's instructions.

Immunoblot analyses of P. gingivalis gingipain and T. denticola dentilisin Immunoblot analyses were performed by mixing the samples at room temperature with Laemmli's sample buffer and heating them at 100°C for 5 minutes prior to electrophoresis. Pre-stained low-range molecular weight SDS-PAGE standards (Bio-Rad) were used as molecular weight markers. For P. gingivalis, gingipain and T. denticola dentilisin served as positive controls. All samples and markers were loaded onto 8% SDS-PAGE gels and electrophoresed at 150 V for one hour. The gels were then transferred onto nitrocellulose membranes, soaked in blocking solution, and incubated overnight with the respective polyclonal anti-gingipain and anti-dentilisin antibodies. Following incubation, the membranes were rinsed four times with TRIS-buffered saline containing 1% Triton X-100, then incubated with antirabbit IgG Horse Radish Peroxidase (HRP) in 5 mL TBST as a secondary antibody and rinsed four times. Detection and development of the immunoblot films were performed in a dark room, with analytes visualized as dark bands on the films. The films were subsequently scanned, and band intensities were quantified using the GS-700 Imaging Densitometer Scanner and the Quantity One program (Bio-Rad).

ELIGIBILITY:
Inclusion Criteria:

* Partially or fully edentulous patients rehabilitated with single or multiple implant-supported prostheses
* Dental implants with functional restorations in place for a minimum of one year, -at least one screw-type titanium implant (single or two-piece) diagnosed with peri-implant mucositis or peri-implantitis and requiring treatment (for diseased groups)
* Non-smokers or former smokers (individuals who had quit smoking for at least five years prior to the study)

Exclusion Criteria:

* Systemic contraindications to dental or surgical treatments
* Active periodontal disease
* Pregnancy or lactation
* Autoimmune or inflammatory diseases
* Uncontrolled diabetes (HbA1c > 7)
* Ongoing corticosteroid therapy
* Current smoking

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Recruitment took place between March 2021 and June 2022, involving patients who attended the clinics of the Department of Periodontology, Sakarya University. These patients were either in the maintenance phase following dental implant therapy, actively undergoing implant treatment, or presenting with complications related to dental implants placed at other centers. A total of 72 participants, encompassing 72 dental implants, were enrolled in the study. These participants were categorized as follows: 23 systemically healthy individuals with peri-implant mucositis, 25 individuals with peri-implantitis, and 24 healthy controls.
Sampling Method: Probability Sample
Enrollment: 72 (Actual)
Dates: Start 2021-03-01 (Actual); Primary Completion 2022-06-01 (Actual); Study Completion 2024-09-01 (Actual)

PRIMARY OUTCOMES:
Bcl-2 family protein levels in peri-implant tissues | From the time of clinical intervention to study completion, an average of 6 months.
  The thawed tissue samples were first weighed and subsequently sectioned into small pieces with disposable scalpels (#11 and #15). The processed tissue fragments were transferred to 2 mL tubes containing four ultrapure zirconium microspheres (3 mm diameter) and 400 μL of lysis buffer. Homogenization was performed using a high-speed tissue homogenizer set at 2000 rpm for four cycles of 60 seconds each, with 20 second intervals on ice to prevent overheating. After homogenization, the samples were centrifuged at 10000 rpm for 4 minutes, and the zirconium beads were removed. Ultrasonication was performed at 0.5 cycle and 100% amplitude in three 5-second cycles, with 20-second intervals on ice between the cycles. The samples were then centrifuged again at 10000 rpm for 4 minutes, and the supernatants were carefully transferred to new tubes.The levels of Bcl-2 family proteins were quantified using a bead-based immunoassay system.

SECONDARY OUTCOMES:
Immunoblot analyses of P. gingivalis gingipain and T. denticola dentilisin | From the time of clinical intervention to study completion, an average of 9 months.
  Immunoblot analyses were performed by mixing the samples at room temperature with Laemmli's sample buffer and heating them at 100°C for 5 minutes prior to electrophoresis. Pre-stained low-range molecular weight SDS-PAGE standards were used as molecular weight markers. For P. gingivalis, gingipain and T. denticola dentilisin served as positive controls. All samples and markers were loaded onto 8% SDS-PAGE gels and electrophoresed at 150 V for one hour. The gels were then transferred onto nitrocellulose membranes, soaked in blocking solution, and incubated overnight with the respective polyclonal anti-gingipain and anti-dentilisin antibodies. Following incubation, the membranes were rinsed four times with TRIS-buffered saline containing 1% Triton X-100, then incubated with antirabbit IgG Horse Radish Peroxidase (HRP) in 5 mL TBST as a secondary antibody and rinsed four times. Detection and development of theimmunoblot films were performed in a dark room.

CONTACTS AND LOCATIONS:
Locations (1):
- Sakarya University, Sakarya, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: Yes
Supporting Information: Study Protocol, SAP, ICF, CSR